CLINICAL TRIAL: NCT02133911
Title: Effects of Ranolazine on Myocardial Perfusion in Patients With Dilated Cardiomyopathy
Brief Title: A Pilot Trial of Ranolazine to Treat Patients With Dilated Cardiomyopathy
Acronym: RAMP-DCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Gregor Poglajen, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHFTX-UMCLJ-1
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controls (No Intervention)
- Ranolazine (Experimental): Initial dose is 375 mg bid. After 2 - 4 weeks the dose is increased to 500 mg bid and after another 2-4 weeks to 750 mg bid. In case of side effects the dose of the drug is to be decreased to the highest dose that the patient is still able to tolerate.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine
  Other Names: Ranexa
  Arms: Ranolazine

SUMMARY:
Recent data suggest that areas of fibrosis and hibernating myocardium develop in patients with non ischemic dilated cardiomyopathy. Ranolazine is a new drug, developed to releave symptoms of angina in patients with stable coronary disease that is not suitable for surgical or percutaneous revascularization. It has been shown that in patients with stable coronary disease Ranolazine improves myocardial perfusion as shown with myocardial nuclear imaging. The aim of this trial is to evaluate effects of ranolazine on myocardial perfusion in patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
Recent data suggest that areas of fibrosis and hibernating myocardium develop in patients with non ischemic dilated cardiomyopathy. Ranolazine is a new drug, developed to releave symptoms of angina in patients with stable coronary disease that is not suitable for surgical or percutaneous revascularization. The main mechanism of action of Ranolazine is the inhibition of late I(Na) thus decreasing the Ca++ load in the cardiomyocites. Consequently oxygen consumption also decreases. It has also been shown that in patients with stable coronary disease Ranolazine improves myocardial perfusion as shown with myocardial nuclear imaging. The aim of this trial is to evaluate effects of ranolazine on myocardial perfusion in patients with dilated cardiomyopathy.

Primary end-point: To determine wheather Ranolazine improves perfusion of the myocardium in patients with non-ischemic dilated cardiomyopathy.

Secondary end-points: To determine wheather Ranolazine improves patients' NYHA functional class, excercise capacity, LV systolic and diastolic function and weather ranolazine affects supraventricular and ventricular arrhythmia occurance/frequency.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of non-ischemic dilated cardiomyopathy
* EF < 35%
* NYHA f.c. II - IV
* Optimal medical management > 6 months
* Age < 75 years and > 18 years

Exclusion Criteria:

* known hypersensitivity to the medication
* age > 75 years or < 18 years
* EF > 35%
* renal insufficiency (GF < 30)
* liver dysfunction (liver tests > 3x the upper normal limit))
* LQT syndrome
* drugs that affect CYP3A4 metabolism (azoles, macrolides, calcineurin inhibitors etc.)
* dementia
* active hemathological or malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05-01; Primary Completion 2015-12-15 (Actual); Study Completion 2016-04-02 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion | 6 months
  To determine wheather Ranolazine improves perfusion of the myocardium in patients with non-ischemic dilated cardiomyopathy assesed by myocardial nuclear imaging.

SECONDARY OUTCOMES:
Excercise capacity | 1, 3 and 6 months
  To determine wheather Ranolazine improves patients' excercise capacity, assesed by 6' walk test
Left ventricular systolic and diastolic function | 1, 3 and 6 months
  To determine wheather Ranolazine improves patients' LV systolic and diastolic function, assesed by LVEF, TDI, LV longitudinal strain and strain rate
Supraventricular and ventricular arrhythmias | 6 months
  To determine wheather Ranolazine affects the occurence of supraventricular and ventricular arrhythmia occurance/frequency using 24 holter monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Poglajen, MD, PhD, Principal Investigator — Advanced Heart Failure and Transplantation Programme, University Medical Center Ljubljana, Slovenia; Bojan Vrtovec, MD, PhD, Study Director — Advanced Heart Failure and Transplantation Programme, University Medical Center Ljubljana, Slovenia
Locations (1):
- Advanced Heart Failure and Transplantation Programme, University Medical Center Ljubljana, Slovenia, Ljubljana, Slovenia